CLINICAL TRIAL: NCT02573584
Title: Vascular Fingerprint to Identify Patients at Risk for Arterial Cardiovascular Events Within the First Year After Start of Cisplatin-based Chemotherapy for Testicular Cancer: a Validation Study
Brief Title: Vascular Fingerprint Validation Study
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201500864
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The vascular fingerprint is a simple selection tool to identify testicular cancer patients with a high risk of arterial cardiovascular events during and in the first year after cisplatin chemotherapy. Eventually, this selection method allows a relative small randomized intervention study with i.e. LMWH during chemotherapy to prove the effectiveness and safety in lowering the chance of an arterial cardiovascular event.

DETAILED DESCRIPTION:
Since the introduction of cisplatin in the late seventies (1), the prognosis of metastatic testicular cancer patients has dramatically improved, with long-term survival rates of 80-90% (2). However, cure rates are compromised by the increased risk of cardiovascular events (3-5). Approximately 1-5% of the patients with metastatic testicular cancer develop arterial cardiovascular events during or shortly after cisplatin- and bleomycin containing chemotherapy (3-7). Arterial cardiovascular events include ischemic stroke and myocardial infarction. These arterial events are a source of serious treatment-induced morbidity and mortality as recently clearly confirmed by Fung (8). No established standard prophylaxis is available. There is an unmet need to have the possibility to identify high risk patients before start of chemotherapy in whom prophylactic anti-coagulant treatment may prevent events (9). An identification tool could maximize the benefit of an intervention without introducing too much unnecessary harm: preventive interventions also carry risk.

Recent data from the investigators' cancer center showed that before chemotherapy 22% of the metastatic cancer patients had ≥3 of the following 5 traditional cardiovascular risk factors present (high risk vascular fingerprint, figure 1): overweight, smoking, hypertension, dyslipidemia and impaired blood glucose. These patients had an increased risk to develop arterial events during or early after chemotherapy: 19% of the patients with a high risk vascular fingerprint developed an arterial cardiovascular event whereas only 2% of the patients with ≤2 risk factors developed an event . The vascular fingerprint seems an easy method to identify which metastatic testicular cancer patients are at a high risk for early arterial events and who may benefit from prophylaxis with for example low molecular weight heparins (LMWHs). To be used in the clinic these data need to be confirmed in an independent cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of metastatic TC and an indication to start with first-line cisplatin-based chemotherapy for metastatic TC
2. Classified into IGCCCG good or intermediate prognosis group
3. Younger than 50 years of age at start of chemotherapy
4. Signed informed consent

Exclusion Criteria:

1. History of previous cardiovascular disease
2. Retroperitoneal mass > 5 cm
3. Indication for anticoagulant therapy at start of chemotherapy

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Newly diagnosed testicular cancer patients before start of chemotherapy.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Development of arterial cardiovascular events | first year after start of chemotherapy
  Primary outcome is development of arterial cardiovascular events within the first year after start of chemotherapy. Events taken into account are: myocardial infarction (WHO ICD-10 I20-I25), ischemic cerebrovascular accidents (WHO ICD-10 I63-I66 and G45) or infarction in other specific organ systems (WHO ICD-10 K76.3, K55, D73.5, M62.2, N28.0)

SECONDARY OUTCOMES:
Overall survival | first year after start of chemotherapy
Response to testicular cancer treatment (no evidence of disease / relapse / no response to treatment) | first year after start of chemotherapy
Development of venous thromboembolic events (VTE) (WHO ICD-10 I26, I80-82) | first year after start of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jourik A Gietema, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (5):
- Netherlands (3):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek ziekenhuis (NKI-AVL), Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - Maastricht University Medical Center (MUMC), Maastricht
- Instituto Portuges de Oncologia Francisco Gentil (IPOLFG), Lisbon, Portugal
- UniversitatsSpital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Einhorn LH, Donohue J. Cis-diamminedichloroplatinum, vinblastine, and bleomycin combination chemotherapy in disseminated testicular cancer. Ann Intern Med. 1977 Sep;87(3):293-8. doi: 10.7326/0003-4819-87-3-293. PMID 71004
- [Result] DeSantis CE, Lin CC, Mariotto AB, Siegel RL, Stein KD, Kramer JL, Alteri R, Robbins AS, Jemal A. Cancer treatment and survivorship statistics, 2014. CA Cancer J Clin. 2014 Jul-Aug;64(4):252-71. doi: 10.3322/caac.21235. Epub 2014 Jun 1. PMID 24890451
- [Result] Weijl NI, Rutten MF, Zwinderman AH, Keizer HJ, Nooy MA, Rosendaal FR, Cleton FJ, Osanto S. Thromboembolic events during chemotherapy for germ cell cancer: a cohort study and review of the literature. J Clin Oncol. 2000 May;18(10):2169-78. doi: 10.1200/JCO.2000.18.10.2169. PMID 10811682
- [Result] Piketty AC, Flechon A, Laplanche A, Nouyrigat E, Droz JP, Theodore C, Fizazi K. The risk of thrombo-embolic events is increased in patients with germ-cell tumours and can be predicted by serum lactate dehydrogenase and body surface area. Br J Cancer. 2005 Oct 17;93(8):909-14. doi: 10.1038/sj.bjc.6602791. PMID 16205699
- [Result] Nuver J, Smit AJ, van der Meer J, van den Berg MP, van der Graaf WT, Meinardi MT, Sleijfer DT, Hoekstra HJ, van Gessel AI, van Roon AM, Gietema JA. Acute chemotherapy-induced cardiovascular changes in patients with testicular cancer. J Clin Oncol. 2005 Dec 20;23(36):9130-7. doi: 10.1200/JCO.2005.01.4092. Epub 2005 Nov 21. PMID 16301596
- [Result] Dieckmann KP, Struss WJ, Budde U. Evidence for acute vascular toxicity of cisplatin-based chemotherapy in patients with germ cell tumour. Anticancer Res. 2011 Dec;31(12):4501-5. PMID 22199322
- [Result] Dieckmann KP, Gerl A, Witt J, Hartmann JT; German Testicular Cancer Study Group. Myocardial infarction and other major vascular events during chemotherapy for testicular cancer. Ann Oncol. 2010 Aug;21(8):1607-1611. doi: 10.1093/annonc/mdp597. Epub 2010 Jan 12. PMID 20067918
- [Result] Fung C, Fossa SD, Milano MT, Sahasrabudhe DM, Peterson DR, Travis LB. Cardiovascular Disease Mortality After Chemotherapy or Surgery for Testicular Nonseminoma: A Population-Based Study. J Clin Oncol. 2015 Oct 1;33(28):3105-15. doi: 10.1200/JCO.2014.60.3654. Epub 2015 Aug 3. PMID 26240226
- [Result] Ramos JD, Yu EY. Cardiovascular Mortality in Testicular Nonseminomatous Germ Cell Tumors: Does Statistical Significance Imply Clinical Significance? J Clin Oncol. 2015 Oct 1;33(28):3075-7. doi: 10.1200/JCO.2015.62.7398. Epub 2015 Aug 24. No abstract available. PMID 26304903
- [Result] Lubberts S, Boer H, Altena R, Meijer C, van Roon AM, Zwart N, Oosting SF, Kamphuisen PW, Nuver J, Smit AJ, Mulder AB, Lefrandt JD, Gietema JA. Vascular fingerprint and vascular damage markers associated with vascular events in testicular cancer patients during and after chemotherapy. Eur J Cancer. 2016 Aug;63:180-8. doi: 10.1016/j.ejca.2016.05.022. Epub 2016 Jun 17. PMID 27322917